CLINICAL TRIAL: NCT01631123
Title: Genetic Determinants of Metabolic Responses to Isocaloric Carbohydrate and Fat Diet Strategies
Brief Title: NUtriGenomic Analysis in Twins
Acronym: NUGAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Charite University, Berlin, Germany (Other); Ernst von Bergmann Hospital (Other); University Hospital Tuebingen (Other); University of Southern California (Other); Ludwig-Maximilians - University of Munich (Other); Heidelberg University (Other); HealthTwist GmbH, Berlin, Germany (Unknown); Max-Planck Institute of Molecular Cell Biology and Genetics (Other); Helmholtz Center Munich (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Chief, Department of Clinical Nutrition, German Institute of Human Nutrition
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BMBF NUGAT 0315424
Record Dates: First submitted 2012-06-01; First posted 2012-06-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Metabolic Response to Dietary Modification
Keywords: Twins; High carbohydrat diet; High fat diet; Isocaloric; Nutrigenomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet interventions (Experimental): Sequential dietary intervention
  Interventions: Other: Isocaloric high carbohydrate diet intervention; Other: Isocaloric high fat diet intervention

INTERVENTIONS:
Other: Isocaloric high carbohydrate diet intervention — Time of 6 week, the last 6 days are standardized
Other: Isocaloric high fat diet intervention — Time of 6 weeks; the first and the last 6 days are standardized

SUMMARY:
This is an intervention study in healthy adult twins with the aim to investigate the genetic determination of metabolic responses towards an isocaloric high carbohydrate, low fat diet versus an isocaloric low carbohydrate, high fat diet.

DETAILED DESCRIPTION:
The impact of carbohydrates, proteins and fatty acids as major components of daily nutrition on the development of metabolic illnesses is an objective of numerous clinical studies. However, the effect of an isocaloric diet on metabolism is less investigated and not well understood. This study aims to reveal genetic determinated metabolic responses to an isocaloric high carbohydrate, low fat diet versus an isocaloric low carbohydrate, high fat diet in healthy twins. This study generates information for further detailed nutrigenomic analysis. Twins receive an isocaloric diet rich in carbohydrates (55% carbohydrates, 15% protein, 30% fat) with dietary counselling for 5 weeks and afterwards with nutrients supplied for 6 days, followed by an isocaloric diet rich in saturated fat (40% carbohydrates, 15% protein, 45% fat) for 6 days with nutrients supplied and for 4 weeks with dietary counselling and again followed by another 6 days when nutrients were supplied. Anthropometry, blood tests and energy expenditure are performed after the period of diet rich in carbohydrates (Carb), after the first 6 days (HFshort) and at the end of the period of diet rich in fat (HFlong).

ELIGIBILITY:
Inclusion Criteria:

* Healthy twins
* BMI 18,5-35kg/m²
* BMI difference < 3kg/m² within the pair of twins
* Stable weight during the last 3 months
* Willingness to comply with the assigned diets over the study period

Exclusion Criteria:

* Consumptive diseases
* Intake of metabolic influence a/o anticoagulent drugs (e.g. cortisone, ASS, antibiotics)
* Diabetes type 1 and type 2
* Pregnancy
* Chronic disease of heart, kidney, liver
* High grade anaemia
* High grade infection disease
* Relevant change of body weight(+/- 2kg)during isoenergetic 12-weeks of dietary intervention
* Missing data about primary outcome measures (IVGTT, MTT, data about dietary intake from food diaries or food protocols)
* Significant deviation from dietary targets during the monitored 12 weeks isoenergetic period
* Allergies including food allergies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Genetic variance of change in insulin secretion and sensitivity after sequential diets | 6,7,12 weeks
  change in insulin secretion and sensitivity measured with an intravenous glucose tolerance test (IVGTT)

SECONDARY OUTCOMES:
Variance of insulin sensitivity after the sequential diets | 6, 7, 12 weeks
  change in insulin sensitivity measured with a meal tolerance test (MTT) allowing for the response of the intestinal hormones
Expression of inflammatory markers in blood and fat tissue | 6,7,12 weeks
  Measurement of gene expression of inflammation cytokines and clock genes
Development of indices for the prediction of fat mass | 6,7,12 weeks
  Change of fat fraction in liver, abdominal and in the total body fat measuring by MRI/H1-spectroscopy, DEXA
Changes in vessel wall thickness of the carotid artery | 6,7,12 weeks
  Vascular ultrasound
Measurement of activity | in the 6th, 7th, 12th week
  each over 6 days measurement: activity protocol, pedometer and activity clock
Detection of the gastric emptying time | 6,7,12 weeks
Assessment of cognitive performance | 0,5,11 weeks
Nutritional and genetic influence on the circadian rhythm | 6, 7, 12 weeks
  measurement of hormones in saliva and urine and of circadian gene expression in monocytes and PBMCs
Epigenetic modification of DNA | 6,7,12 weeks
  Change in adipose tissue DNA methylation pattern
Biometric data | 6,7,12 weeks
  Nutritional impact of the blood pressure, weight, body mass index, waist-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof, Principal Investigator — German Institute of Human Nutrition Potsdam-Rehbruecke
Locations (1):
- German Institute of Human Nutrition, Potsdam-Rehbruecke, Nuthetal, Germany

REFERENCES:
- [Derived] Schuler R, Seebeck N, Osterhoff MA, Witte V, Floel A, Busjahn A, Jais A, Bruning JC, Frahnow T, Kabisch S, Pivovarova O, Hornemann S, Kruse M, Pfeiffer AFH. VEGF and GLUT1 are highly heritable, inversely correlated and affected by dietary fat intake: Consequences for cognitive function in humans. Mol Metab. 2018 May;11:129-136. doi: 10.1016/j.molmet.2018.02.004. Epub 2018 Feb 12. PMID 29506909
- [Derived] Schuler R, Osterhoff MA, Frahnow T, Seltmann AC, Busjahn A, Kabisch S, Xu L, Mosig AS, Spranger J, Mohlig M, Hornemann S, Kruse M, Pfeiffer AF. High-Saturated-Fat Diet Increases Circulating Angiotensin-Converting Enzyme, Which Is Enhanced by the rs4343 Polymorphism Defining Persons at Risk of Nutrient-Dependent Increases of Blood Pressure. J Am Heart Assoc. 2017 Jan 17;6(1):e004465. doi: 10.1161/JAHA.116.004465. PMID 28096099
- [Derived] Pivovarova O, Jurchott K, Rudovich N, Hornemann S, Ye L, Mockel S, Murahovschi V, Kessler K, Seltmann AC, Maser-Gluth C, Mazuch J, Kruse M, Busjahn A, Kramer A, Pfeiffer AF. Changes of Dietary Fat and Carbohydrate Content Alter Central and Peripheral Clock in Humans. J Clin Endocrinol Metab. 2015 Jun;100(6):2291-302. doi: 10.1210/jc.2014-3868. Epub 2015 Mar 30. PMID 25822100